CLINICAL TRIAL: NCT05870956
Title: Economic Burden Associated With Nintedanib Non-adherence Among Medicare Beneficiaries With IPF
Brief Title: Burden of Nintedanib Non-adherence Among Idiopathic Pulmonary Fibrosis (IPF) Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0520
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (5):
- High nintedanib adherence: Community-dwelling Idiopathic Pulmonary Fibrosis (IPF) patients with 66 years of age or older at the time of the first nintedanib prescription (between 01-Oct-2014 and 31-Oct-2018), and continuous Medicare hospital (Part A), physician (Part B) and pharmacy (Part D) coverage (between 01-Oct-2013 to 31-12-2020). Patients in high adherence group presented a mean adherence estimate of 0.96 (proportion of days covered - PDC) in a period of 12 months after nintedanib first initiation.
  Interventions: Drug: Nintedanib
- Moderate nintedanib adherence: Community-dwelling Idiopathic Pulmonary Fibrosis (IPF) patients with 66 years of age or older at the time of the first nintedanib prescription (between 01-Oct-2014 and 31-Oct-2018), and continuous Medicare hospital (Part A), physician (Part B) and pharmacy (Part D) coverage (between 01-Oct-2013 to 31-12-2020). Patients in moderate adherence group presented a mean adherence estimate of 0.71 (proportion of days covered - PDC) in a period of 12 months after nintedanib first initiation.
  Interventions: Drug: Nintedanib
- High-then-poor nintedanib adherence: Community-dwelling Idiopathic Pulmonary Fibrosis (IPF) patients with 66 years of age or older at the time of the first nintedanib prescription (between 01-Oct-2014 and 31-Oct-2018), and continuous Medicare hospital (Part A), physician (Part B) and pharmacy (Part D) coverage (between 01-Oct-2013 to 31-12-2020). Patients in high-then-poor adherence group presented a mean adherence estimate of 0.74 (proportion of days covered - PDC) in a period of 12 months after nintedanib first initiation, with a high adherence in the first 7 months followed by a sharp decline.
  Interventions: Drug: Nintedanib
- Delayed-poor nintedanib adherence: Community-dwelling Idiopathic Pulmonary Fibrosis (IPF) patients with 66 years of age or older at the time of the first nintedanib prescription (between 01-Oct-2014 and 31-Oct-2018), and continuous Medicare hospital (Part A), physician (Part B) and pharmacy (Part D) coverage (between 01-Oct-2013 to 31-12-2020). Patients in delayed poor adherence group presented a mean adherence estimate of 0.36 (proportion of days covered - PDC) in a period of 12 months after nintedanib first initiation, with a high adherence in the first 2 months followed by a constant decline.
  Interventions: Drug: Nintedanib
- Early-poor nintedanib adherence: Community-dwelling Idiopathic Pulmonary Fibrosis (IPF) patients with 66 years of age or older at the time of the first nintedanib prescription (between 01-Oct-2014 and 31-Oct-2018), and continuous Medicare hospital (Part A), physician (Part B) and pharmacy (Part D) coverage (between 01-Oct-2013 to 31-12-2020). Patients in early-poor adherence group presented a mean adherence estimate of 0.13 (proportion of days covered - PDC) in a period of 12 months after nintedanib first initiation, with a high adherence in the first month followed by a sharp decline.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib
  Other Names: Ofev®

SUMMARY:
This study has two objectives:

1. To assess the association between nintedanib adherence trajectory group (as measured from a Group-based Trajectory Modelling (GBTM)) and health care resource use, with a focus on inpatient hospitalization, among patients with Idiopathic Pulmonary Fibrosis (IPF).
2. To assess the association between a patient's nintedanib adherence trajectory group (as measured from a GBTM) and their medical costs among patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

* Newly initiated nintedanib during 10/01/2014 to 12/31/2018
* Were at least 66 years old as of the date of their first nintedanib prescription claim (index date)
* Qualified for Medicare based on age
* Had at least 12 months of continuous enrollment in Medicare Parts A, B and D before (baseline period) and 12 months after the index date (follow-up period)
* Had at least one inpatient or two outpatient claims (>14 days apart) with a diagnosis code for IPF (ICD-10-CM: J84.112; ICD-9-CM: 516.31) during the baseline period

Exclusion Criteria:

* Had any history of pirfenidone or nintedanib use during the baseline period
* Had any history of lung transplant during the baseline, index date or follow-up periods
* Had any claims for skilled nursing facility, long-term care facility or hospice during the baseline, index date or follow-up period
* Had evidence (≥2 ICD-9-CM or ICD-10-CM diagnosis codes on different dates) during the baseline period of any of the following conditions: lung cancer, autoimmune, or connective tissue diseases (i.e., rheumatoid arthritis (RA), sarcoidosis, systemic lupus erythematosus (SLE), dermatopolymyositis, systemic sclerosis, Sjogren's, and mixed connective tissue disease (CTD)) during the baseline period
* Had dual eligibility of Medicare and Medicaid
* Had history of using pirfenidone at the same time with nintedanib during follow-up

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: IPF patients in United States which were newly initiated on nintedanib during 10-Jan-2014 to 31-Dec-2018.
Sampling Method: Non-Probability Sample
Enrollment: 1798 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medicus Economics, LCC, Milton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective cohort study using United States (US) Medicare hospital (Part A), physician (Part B) and pharmacy (Part D) administrative claims to characterize the trajectory of adherence to nintedanib in Idiopathic Pulmonary Fibrosis (IPF) patients as measured during the first year following initiation. The study uses data covering the period of 01-Oct-2013 to 31-12-2020, capturing the first use of nintedanib (index date) between 01-Oct-2014 and 31-Oct-2018.
Pre-assignment Details: Patients that met all inclusion criteria and none of the exclusion criteria were followed 12 months before the first use of nintedanib (baseline period) to 24 months after its initiation.
Period: Overall Study
Arm/Group | High Nintedanib Adherence | Moderate Nintedanib Adherence | High-then-poor Nintedanib Adherence | Delayed-poor Nintedanib Adherence | Early-poor Nintedanib Adherence
Started | 781 | 202 | 190 | 255 | 370
Completed | 781 | 202 | 190 | 255 | 370
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: Community-dwelling Idiopathic Pulmonary Fibrosis (IPF) patients with Medicare hospital, physician and pharmacy coverage data, between 01-Oct-2013 to 31-12-2020, who met all inclusion criteria and none of the exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Nintedanib Adherence | Moderate Nintedanib Adherence | High-then-poor Nintedanib Adherence | Delayed-poor Nintedanib Adherence | Early-poor Nintedanib Adherence | Total
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370 | 1798
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.65 (5.36) | 75.21 (5.45) | 75.89 (5.60) | 76.29 (5.61) | 76.21 (5.62) | 75.40 (5.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 89 | 66 | 117 | 177 | 700
  Male | 530 | 113 | 124 | 138 | 193 | 1098
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-hispanic white | 718 | 183 | 171 | 237 | 329 | 1638
  Not non-hispanic white | 63 | 19 | 19 | 18 | 41 | 160

OUTCOME MEASURES:

1. Primary Outcome: Total All-cause Medical Costs
Description: Total all-cause medical costs per patient calculated as the sum of the total amounts paid for all medical services by the payer and the patient. The types of medical services covered by Medicare included inpatient facility, outpatient facility, skilled nursing facility, home health care, hospice, durable medical equipment, clinician office visits, and other physician services covered under the Part B benefit. The costs with prescriptions covered under Part D benefit were excluded from this outcome analysis.
Time Frame: At day 360 after the index date, i.e., between 01-Oct-2014 and 31-Oct-2018.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | High Nintedanib Adherence | Moderate Nintedanib Adherence | High-then-poor Nintedanib Adherence | Delayed-poor Nintedanib Adherence | Early-poor Nintedanib Adherence
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States dollars | 12647.73 (16996) | 13580.61 (18479) | 17549.74 (27854) | 15375.10 (16999) | 18110.14 (26365)
Statistical Analysis 1: Comparison: High Nintedanib Adherence vs Moderate Nintedanib Adherence; Test type: Other; p = 0.516, ANOVA; Mean Difference (Net) = 932.88, 95% CI 2-sided [-1880.17 to 3745.94] — The net difference was calculated as: Comparator - Reference where High nintedanib adherence group was used as reference
Statistical Analysis 2: Comparison: High Nintedanib Adherence vs High-then-poor Nintedanib Adherence; Test type: Other; p = 0.020, ANOVA; Mean Difference (Net) = 4902.02, 95% CI 2-sided [767.60 to 9036.43] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: High Nintedanib Adherence vs Delayed-poor Nintedanib Adherence; Test type: Other; p = 0.026, ANOVA; Mean Difference (Net) = 2727.38, 95% CI 2-sided [323.48 to 5131.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: High Nintedanib Adherence vs Early-poor Nintedanib Adherence; Test type: Other; p = 0.000, ANOVA; Mean Difference (Net) = 5462.41, 95% CI 2-sided [2520.93 to 8403.90] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Total IPF-related Medical Costs
Description: The total Idiopathic Pulmonary Fibrosis (IPF) related medical costs per patient were calculated as the sum of the total amounts paid by the payers and the patients for all medical services for an IPF-related reason containing at least one IPF diagnosis code.
Time Frame: At year 1 after the index date, i.e., between 01-Oct-2014 and 31-Oct-2018.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | High Nintedanib Adherence | Moderate Nintedanib Adherence | High-then-poor Nintedanib Adherence | Delayed-poor Nintedanib Adherence | Early-poor Nintedanib Adherence
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States dollars | 3239.75 (6313) | 2935.82 (4574) | 6011.81 (16239) | 3696.54 (6525) | 3860.62 (12947)
Statistical Analysis 1: Comparison: High Nintedanib Adherence vs Moderate Nintedanib Adherence; Test type: Other; p = 0.439, ANOVA; Mean Difference (Net) = -303.94, 95% CI 2-sided [-1074.77 to 466.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: High Nintedanib Adherence vs High-then-poor Nintedanib Adherence; Test type: Other; p = 0.021, ANOVA; Mean Difference (Net) = 2772.06, 95% CI 2-sided [422.10 to 5122.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: High Nintedanib Adherence vs Delayed-poor Nintedanib Adherence; Test type: Other; p = 0.328, ANOVA; Mean Difference (Net) = 456.79, 95% CI 2-sided [-458.64 to 1372.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: High Nintedanib Adherence vs Early-poor Nintedanib Adherence; Test type: Other; p = 0.382, ANOVA; Mean Difference (Net) = 620.87, 95% CI 2-sided [-771.77 to 2013.51] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: All-cause Inpatient Hospitalization
Description: Percentage of patients with at least one inpatient hospitalization for any cause in the first year of nintedanib initiation. Percentages were rounded to one decimal place.
Time Frame: At year 1 after the index date, i.e., between 01-Oct-2014 and 31-Oct-2018.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | High Nintedanib Adherence | Moderate Nintedanib Adherence | High-then-poor Nintedanib Adherence | Delayed-poor Nintedanib Adherence | Early-poor Nintedanib Adherence
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Percentage of participants | 20.4 | 22.8 | 30.0 | 29.4 | 26.8
Statistical Analysis 1: Comparison: High Nintedanib Adherence vs Moderate Nintedanib Adherence; Test type: Other; p = 0.463, Chi-squared; Mean Difference (Net) = 2.4, 95% CI 2-sided [-4.0 to 8.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: High Nintedanib Adherence vs High-then-poor Nintedanib Adherence; Test type: Other; p = 0.008, Chi-squared; Mean Difference (Net) = 9.6, 95% CI 2-sided [2.5 to 16.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: High Nintedanib Adherence vs Delayed-poor Nintedanib Adherence; Test type: Other; p = 0.005, Chi-squared; Mean Difference (Net) = 9.1, 95% CI 2-sided [2.8 to 15.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: High Nintedanib Adherence vs Early-poor Nintedanib Adherence; Test type: Other; p = 0.019, Chi-squared; Mean Difference (Net) = 6.4, 95% CI 2-sided [1.1 to 11.7] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: IPF-related Inpatient Hospitalization
Description: Percentage of patients with at least one inpatient hospitalization for any Idiopathic Pulmonary Fibrosis (IPF)-related cause in the first year of nintedanib initiation. Percentages were rounded to one decimal place.
Time Frame: At year 1 after the index date, i.e., between 01-Oct-2014 and 31-Oct-2018.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | High Nintedanib Adherence | Moderate Nintedanib Adherence | High-then-poor Nintedanib Adherence | Delayed-poor Nintedanib Adherence | Early-poor Nintedanib Adherence
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Percentage of participants | 10.8 | 11.4 | 19.5 | 14.1 | 12.2
Statistical Analysis 1: Comparison: High Nintedanib Adherence vs Moderate Nintedanib Adherence; Test type: Other; p = 0.801, Chi-squared; Mean Difference (Net) = 0.6, 95% CI 2-sided [-4.3 to 5.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: High Nintedanib Adherence vs High-then-poor Nintedanib Adherence; Test type: Other; p = 0.005, Chi-squared; Mean Difference (Net) = 8.7, 95% CI 2-sided [2.7 to 14.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: High Nintedanib Adherence vs Delayed-poor Nintedanib Adherence; Test type: Other; p = 0.170, Chi-squared; Mean Difference (Net) = 3.4, 95% CI 2-sided [-1.4 to 8.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: High Nintedanib Adherence vs Early-poor Nintedanib Adherence; Test type: Other; p = 0.489, Chi-squared; Mean Difference (Net) = 1.4, 95% CI 2-sided [-2.6 to 5.4] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: As this is a non-interventional study with secondary use of data retrieved from Medicare administrative claims, safety monitoring and safety reporting on an individual case level is not applicable. All-Cause Mortality, Serious Adverse Events and Other Adverse Events are not collected in the database. "0" total Number of Participants at Risk means "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | High Nintedanib Adherence | Moderate Nintedanib Adherence | High-then-poor Nintedanib Adherence | Delayed-poor Nintedanib Adherence | Early-poor Nintedanib Adherence
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study limitations included: the data source was composed of administrative claims; the adherence exposure was based on prescription fill data; the outcomes were measured contemporaneously with nintedanib adherence; the outcomes consisted of inpatient hospitalization and total medical spending; the early-poor adherence group consisted of a smaller sample; sample selection bias due to the time frame chosen for patient selection; COVID-19 might have impacted health care consumption patterns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT05870956/Prot_SAP_000.pdf